CLINICAL TRIAL: NCT05454683
Title: Effect of Melatonin Plus Zinc Supplementation on Fatigue, Pain, Sleep Disturbances, Anxiety and Depression, and Autonomic Dysfunction in ME/CFS: a Randomized, Double-blind, Placebo-controlled Study
Brief Title: Melatonin and Zinc Administration on Cardinal Symptoms in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome
Acronym: MelatoZincME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratorios Viñas, S.A. (Industry)
Collaborators: Laboratorio Echevarne (Industry); Hospital Vall d'Hebron (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IC/LV/MEL-ZN/SFC2
Record Dates: First submitted 2022-06-30; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Chronic Fatigue Syndrome; Myalgic Encephalomyelitis
Keywords: melatonin; zinc; fatigue; sleep quality; quality of life; pain; anxiety and depression; actigraphy; heart rate variability; orthostatic intolerance
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Fatigue; Sleep Initiation and Maintenance Disorders; Pain; Anxiety Disorders; Depression; Orthostatic Intolerance | interventions — Melatonin; Zinc; Isomaltose; stearic acid; Excipients

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin plus Zinc (Experimental): Dietary Supplement:
  53 patients treated with melatonin 1 mg plus Zinc 10 mg
  Interventions: Dietary Supplement: melatonin plus zinc
- Placebo (Placebo Comparator): 53 patients treated with isomaltose and magnesium stearate (excipients)
  Interventions: Other: isomaltose and magnesium stearate

INTERVENTIONS:
Dietary Supplement: melatonin plus zinc — One capsule with melatonin 1mg plus zinc 10 mg o.d. 30 minutes before bedtime, at least 1 hour after dinner during 4 months
  Other Names: MelatoZinc
  Arms: Melatonin plus Zinc
Other: isomaltose and magnesium stearate — One capsule with excipients o.d. 30 minutes before bedtime, at least 1 hour after dinner during 4 months
  Other Names: excipients
  Arms: Placebo

SUMMARY:
The aim of the study is to investigate the effects of oral melatonin and zinc supplementation on core features in individuals with ME/CFS

DETAILED DESCRIPTION:
Myalgic Encephalomyelitis, also known as Chronic Fatigue Syndrome (ME/CFS) is a heterogeneous condition characterized mainly by debilitating and prolonged fatigue, post-exertional malaise (physical, mental and emotional), unrefreshing sleep, cognitive impairment, and orthostatic intolerance with prolonged recovery that is not relieved by rest. Currently, the etiopathogenic mechanisms of ME/CFS are unknown. At present, there is no diagnostic test or effective treatment. MelatoZinc is a food supplement composed of melatonin and zinc, which could contribute to the circadian rhythm homeostasis and regulation of redox imbalance and immune response.

The aim is to evaluate the efficacy and safety of oral treatment with MelatoZinc on the symptomatic complex of fatigue in a larger Spanish ME/CFS population.

This is a single-center, randomized, double-blind, placebo controlled clinical trial. It will include a total of 106 ME/CFS patients who met 2011 ICC criteria for ME/CFS. All patients will take one capsule daily for 16 weeks. Group A will receive MelatoZinc (1 mg melatonin plus 10 mg zinc), and group B will receive a placebo (excipients: isomaltose and magnesium stearate). Clinical symptoms will be evaluated, and standardized questionnaires will be applied to assess the impact of fatigue, pain, anxiety-depression symptoms, sleep quality, dysautonomia, and quality of life. Heart rate variability (HRV) and orthostatic intolerance (10-min NASA Lean Test) will be performed to evaluate autonomic dysfunction. Sleep efficiency will be estimated through an actigraph sensor

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18 and 65 years of age.
2. Patients with ME/CFS who met the diagnostic criteria (2011 ICC criteria) from the Central Sensitization Syndrome Unit (USSC) at the Vall d'Hebron University Hospital.
3. Patients who freely give written consent.

Exclusion Criteria:

1. Any active medical condition that explained chronic fatigue (untreated hypothyroidism, sleep apnea, narcolepsy, medication side-effects).
2. Previous diagnosis not unequivocally resolved (chronic hepatitis, malignancy).
3. Past or current psychiatric disorders (major depressive disorder with psychotic or melancholic features, bipolar disorder, schizophrenia, delusional disorder, dementias, anorexia nervosa, bulimia nervosa).
4. Participation in another clinical trial of the same or different nature in the 30 days prior to study inclusion.
5. In the judgment of the investigator, inability to follow the instructions or to complete the treatment satisfactorily.
6. Failure to provide signed informed consent.
7. Current consumption of medications that may interfere with the results and/or whose withdrawal may be a relevant problem.
8. Anticoagulant treatment.
9. Pregnancy or breast-feeding, or had not used oral contraceptives or other hormonal preparations in the previous 6 months.
10. Smoking, alcohol intake or substance abuse.
11. Severe obesity (class 3 BMI ≥ 40 kg/m2).
12. Hypersensitivity to melatonin and/or zinc dietary supplements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2022-09-05 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-reported fatigue as assessed by the 40-item Fatigue Impact Scale (FIS-40) over the baseline in the study participants. | During 4 months of treatment and 8 weeks after discontinuation of dietary therapy
  The FIS-40 includes three subscales of the perceived impact of fatigue: cognitive (10 items), physical (10 items) and psychosocial functions (20 items), each item being scored from 0 (no fatigue) to 4 (severe fatigue). The total score is calculated by adding together the responses from the 40 questions (range 0-160). Higher scores indicate more functional limitations due to fatigue.

SECONDARY OUTCOMES:
The health-related quality of life (HRQoL) as assessed by the Short-Form 36-Item Health Survey (SF-36) over the baseline in the study participants. | During 4 months of treatment and 8 weeks after discontinuation of dietary therapy
  The SF-36 is a broadly-based self-reported survey on health-related physical and mental functioning status. It assesses functioning on eight subscales, including domains of physical functioning, physical role, bodily pain, general health, social functioning, vitality, emotional role and mental health, and two general subscales covering the physical and mental health domains on a 0-100 score. Lower scores indicate a more negative impact of an individual's health on functioning.
Sleep disturbances as assessed by the Pittsburgh Sleep Quality Index (PSQI) questionnaire over the baseline in the study participants. | During 4 months of treatment and 8 weeks after discontinuation of dietary therapy
  The PSQI is the self-administered 19-item questionnaire. PSQI scores are obtained on each of seven components of sleep quality: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep perturbations, use of sleeping medication and daytime dysfunction. Each item is scored from 0 to 3 (0 = no sleep problems and 3 = severe sleep problems). The global PSQI score ranges from 0 to 21 points, with scores of >5 indicating poorer sleep quality.
Sleepiness as assessed by the Epworth Sleepiness Scale (ESS) over the baseline in the study participants. | During 4 months of treatment and 8 weeks after discontinuation of dietary therapy
  The ESS is a short, self-administered questionnaire that consists of eight questions asking to rate how likely it is to fall asleep in everyday situations (each question can be scored from 0 to 3 points: '0' indicates no sleepiness, and '3' indicates significant sleepiness). It provides a total score which has been shown to relate to the subject's level of daytime sleepiness (total score is ranging from 0 to 24 points).
Sleep latency as assessed by an actigraph sensor over the baseline in the study participants. | During 4 months of treatment and 8 weeks after discontinuation of dietary therapy
  An actigraph (Actiwatch Spectrum Plus® from Philips Respironics, Linton Instrumentation, UK) on the wrist of the non-dominant arm is continuously recording for seven days. The same device was programmed to collect data on motor activity (accelerometer) and light type/intensity (lux) at one minute intervals. These variables were recorded and stored in the device's memory for data analysis.
Sleep onset as assessed by an actigraph sensor over the baseline in the study participants | During 4 months of treatment and 8 weeks after discontinuation of dietary therapy
  An actigraph (Actiwatch Spectrum Plus® from Philips Respironics, Linton Instrumentation, UK) on the wrist of the non-dominant arm is continuously recording for seven days. The same device is programmed to collect data on motor activity (accelerometer) and light type/intensity (lux) at one minute intervals. These variables will be recorded and stored in the device's memory for further data analysis.
Sleep efficiency as assessed by an actigraph sensor over the baseline in the study participants. | During 4 months of treatment and 8 weeks after discontinuation of dietary therapy
  An actigraph (Actiwatch Spectrum Plus® from Philips Respironics, Linton Instrumentation, UK) on the wrist of the non-dominant arm is continuously recording for seven days. The same device is programmed to collect data on motor activity (accelerometer) and light type/intensity (lux) at one minute intervals. These variables will be recorded and stored in the device's memory for further data analysis.
Total sleep time as assessed by an actigraph sensor over the baseline in the study participants. | During 4 months of treatment and 8 weeks after discontinuation of dietary therapy
  An actigraph (Actiwatch Spectrum Plus® from Philips Respironics, Linton Instrumentation, UK) on the wrist of the non-dominant arm is continuously recording for seven days. The same device is programmed to collect data on motor activity (accelerometer) and light type/intensity (lux) at one minute intervals. These variables will be recorded and stored in the device's memory for further data analysis.
Wake time as assessed by an actigraph sensor over the baseline in the study participants. | During 4 months of treatment and 8 weeks after discontinuation of dietary therapy
  An actigraph (Actiwatch Spectrum Plus® from Philips Respironics, Linton Instrumentation, UK) on the wrist of the non-dominant arm is continuously recording for seven days. The same device is programmed to collect data on motor activity (accelerometer) and light type/intensity (lux) at one minute intervals. These variables will be recorded and stored in the device's memory for further data analysis.
Number of awakenings as assessed by an actigraph sensor over the baseline in the study participants. | During 4 months of treatment and 8 weeks after discontinuation of dietary therapy
  An actigraph (Actiwatch Spectrum Plus® from Philips Respironics, Linton Instrumentation, UK) on the wrist of the non-dominant arm is continuously recording for seven days. The same device is programmed to collect data on motor activity (accelerometer) and light type/intensity (lux) at one minute intervals. These variables will be recorded and stored in the device's memory for further data analysis.
Heart rate variability (HRV) as recorded by the FitLab software over the baseline in the study participants. | During 4 months of treatment and 8 weeks after discontinuation of dietary therapy
  Changes in the cardiovagal autonomic dysfuntion will be continuously assessed and recorded for the R-R intervals over 5-min periods at rest and in the supine position on different days using the FitLab software.
Orthostatic intolerance as assessed by the active standing test (10-minute NASA Lean test) over the baseline in the study participants. | During 4 months of treatment and 8 weeks after discontinuation of dietary therapy
  The 10-minute NLT is a well-established non-invasive procedure used to assess impaired cardiovascular responses to standing and to diagnose OI phenotypes. It records objective hemodynamic parameters (blood pressure and heart rate). The participants will be first asked to lie down during 5 minutes and then to stand and lean against a wall, with heels 6-8 inches from the wall. Throughout the recording, participants will be asked to remain motionless, quiet and any talking or movement will be discouraged, except for reporting any symptoms of concern.
Pain intensity as assessed by a visual analog scale (VAS) over the baseline in the study participants. | During 4 months of treatment and 8 weeks after discontinuation of dietary therapy
  The pain VAS is a continuous and unidimensional measure of pain intensity. It comprised of a horizontal line of 10-centimeters in length, anchored by 2 verbal descriptors, one for each symptom extreme. "No pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain"(score of 10).
Anxiety and depression symptoms as assessed by the Hospital Anxiety and Depression Scale (HADS) over the baseline in the study participants. | During 4 months of treatment and 8 weeks after discontinuation of dietary therapy
  The HADS is a validated self-reported tool composed of 14 items (seven related to anxiety symptoms and seven to depression). Each item is scored from 0-3, and thus, scores range from 0 to 21; scores of 0-7 are interpreted as normal, 8-10 as mild, 11-14 as moderate, and 15-21 as severe for either anxiety or depression. The total HADS score ranges from 0 (no anxiety or depression) to 42 (severe anxiety and depression).
Side effect of treatment | During 4 months of treatment and 8 weeks after discontinuation of dietary therapy
  Treatment side effects will be collected from each participant during clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: José Alegre, MD, PhD, Principal Investigator — Vall d'Hebron University Hospital
Locations (1):
- Vall d'Hebron University Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castro-Marrero J, Zaragoza MC, Lopez-Vilchez I, Galmes JL, Cordobilla B, Maurel S, Domingo JC, Alegre-Martin J. Effect of Melatonin Plus Zinc Supplementation on Fatigue Perception in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome: A Randomized, Double-Blind, Placebo-Controlled Trial. Antioxidants (Basel). 2021 Jun 23;10(7):1010. doi: 10.3390/antiox10071010. PMID 34201806
- [Background] Castro-Marrero J, Domingo JC, Cordobilla B, Ferrer R, Giralt M, Sanmartin-Sentanes R, Alegre-Martin J. Does Coenzyme Q10 Plus Selenium Supplementation Ameliorate Clinical Outcomes by Modulating Oxidative Stress and Inflammation in Individuals with Myalgic Encephalomyelitis/Chronic Fatigue Syndrome? Antioxid Redox Signal. 2022 Apr;36(10-12):729-739. doi: 10.1089/ars.2022.0018. PMID 35229657
- [Background] Castro-Marrero J, Zacares M, Almenar-Perez E, Alegre-Martin J, Oltra E. Complement Component C1q as a Potential Diagnostic Tool for Myalgic Encephalomyelitis/Chronic Fatigue Syndrome Subtyping. J Clin Med. 2021 Sep 15;10(18):4171. doi: 10.3390/jcm10184171. PMID 34575280
- [Background] Castro-Marrero J, Segundo MJ, Lacasa M, Martinez-Martinez A, Sentanes RS, Alegre-Martin J. Effect of Dietary Coenzyme Q10 Plus NADH Supplementation on Fatigue Perception and Health-Related Quality of Life in Individuals with Myalgic Encephalomyelitis/Chronic Fatigue Syndrome: A Prospective, Randomized, Double-Blind, Placebo-Controlled Trial. Nutrients. 2021 Jul 30;13(8):2658. doi: 10.3390/nu13082658. PMID 34444817
- [Background] Baklund IH, Dammen T, Moum TA, Kristiansen W, Duarte DS, Castro-Marrero J, Helland IB, Strand EB. Evaluating Routine Blood Tests According to Clinical Symptoms and Diagnostic Criteria in Individuals with Myalgic Encephalomyelitis/Chronic Fatigue Syndrome. J Clin Med. 2021 Jul 14;10(14):3105. doi: 10.3390/jcm10143105. PMID 34300271
- [Background] Capdevila L, Castro-Marrero J, Alegre J, Ramos-Castro J, Escorihuela RM. Analysis of Gender Differences in HRV of Patients with Myalgic Encephalomyelitis/Chronic Fatigue Syndrome Using Mobile-Health Technology. Sensors (Basel). 2021 May 28;21(11):3746. doi: 10.3390/s21113746. PMID 34071326
- [Background] Domingo JC, Cordobilla B, Ferrer R, Giralt M, Alegre-Martin J, Castro-Marrero J. Are Circulating Fibroblast Growth Factor 21 and N-Terminal Prohormone of Brain Natriuretic Peptide Promising Novel Biomarkers in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome? Antioxid Redox Signal. 2021 Jun 20;34(18):1420-1427. doi: 10.1089/ars.2020.8230. Epub 2021 Feb 11. PMID 33353469
- [Background] Gomez-Mora E, Carrillo J, Urrea V, Rigau J, Alegre J, Cabrera C, Oltra E, Castro-Marrero J, Blanco J. Impact of Long-Term Cryopreservation on Blood Immune Cell Markers in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome: Implications for Biomarker Discovery. Front Immunol. 2020 Nov 17;11:582330. doi: 10.3389/fimmu.2020.582330. eCollection 2020. PMID 33329554
- [Background] Giloteaux L, O'Neal A, Castro-Marrero J, Levine SM, Hanson MR. Cytokine profiling of extracellular vesicles isolated from plasma in myalgic encephalomyelitis/chronic fatigue syndrome: a pilot study. J Transl Med. 2020 Oct 12;18(1):387. doi: 10.1186/s12967-020-02560-0. PMID 33046133
- [Background] Estevez-Lopez F, Mudie K, Wang-Steverding X, Bakken IJ, Ivanovs A, Castro-Marrero J, Nacul L, Alegre J, Zalewski P, Slomko J, Strand EB, Pheby D, Shikova E, Lorusso L, Capelli E, Sekulic S, Scheibenbogen C, Sepulveda N, Murovska M, Lacerda E. Systematic Review of the Epidemiological Burden of Myalgic Encephalomyelitis/Chronic Fatigue Syndrome Across Europe: Current Evidence and EUROMENE Research Recommendations for Epidemiology. J Clin Med. 2020 May 21;9(5):1557. doi: 10.3390/jcm9051557. PMID 32455633
- [Background] Cheema AK, Sarria L, Bekheit M, Collado F, Almenar-Perez E, Martin-Martinez E, Alegre J, Castro-Marrero J, Fletcher MA, Klimas NG, Oltra E, Nathanson L. Unravelling myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS): Gender-specific changes in the microRNA expression profiling in ME/CFS. J Cell Mol Med. 2020 May;24(10):5865-5877. doi: 10.1111/jcmm.15260. Epub 2020 Apr 14. PMID 32291908
- [Background] Escorihuela RM, Capdevila L, Castro JR, Zaragoza MC, Maurel S, Alegre J, Castro-Marrero J. Reduced heart rate variability predicts fatigue severity in individuals with chronic fatigue syndrome/myalgic encephalomyelitis. J Transl Med. 2020 Jan 6;18(1):4. doi: 10.1186/s12967-019-02184-z. PMID 31906988
- [Background] Bhatia S, Olczyk N, Jason LA, Alegre J, Fuentes-Llanos J, Castro-Marrero J. A Cross-National Comparison of Myalgic Encephalomyelitis and Chronic Fatigue Syndrome at Tertiary Care Settings from the US and Spain. Am J Soc Sci Humanit. 2020;5(1):104-115. doi: 10.20448/801.51.104.115. Epub 2019 Dec 19. PMID 34109300
- [Background] Castro-Marrero J, Faro M, Zaragoza MC, Aliste L, de Sevilla TF, Alegre J. Unemployment and work disability in individuals with chronic fatigue syndrome/myalgic encephalomyelitis: a community-based cross-sectional study from Spain. BMC Public Health. 2019 Jun 28;19(1):840. doi: 10.1186/s12889-019-7225-z. PMID 31253111
- [Background] Estevez-Lopez F, Castro-Marrero J, Wang X, Bakken IJ, Ivanovs A, Nacul L, Sepulveda N, Strand EB, Pheby D, Alegre J, Scheibenbogen C, Shikova E, Lorusso L, Capelli E, Sekulic S, Lacerda E, Murovska M; European Network on ME/CFS (EUROMENE). Prevalence and incidence of myalgic encephalomyelitis/chronic fatigue syndrome in Europe-the Euro-epiME study from the European network EUROMENE: a protocol for a systematic review. BMJ Open. 2018 Sep 4;8(9):e020817. doi: 10.1136/bmjopen-2017-020817. PMID 30181183
- [Background] Cambras T, Castro-Marrero J, Zaragoza MC, Diez-Noguera A, Alegre J. Circadian rhythm abnormalities and autonomic dysfunction in patients with Chronic Fatigue Syndrome/Myalgic Encephalomyelitis. PLoS One. 2018 Jun 6;13(6):e0198106. doi: 10.1371/journal.pone.0198106. eCollection 2018. PMID 29874259
- [Background] Castro-Marrero J, Zaragoza MC, Gonzalez-Garcia S, Aliste L, Saez-Francas N, Romero O, Ferre A, Fernandez de Sevilla T, Alegre J. Poor self-reported sleep quality and health-related quality of life in patients with chronic fatigue syndrome/myalgic encephalomyelitis. J Sleep Res. 2018 Dec;27(6):e12703. doi: 10.1111/jsr.12703. Epub 2018 May 16. PMID 29770505
- [Background] Castro-Marrero J, Serrano-Pertierra E, Oliveira-Rodriguez M, Zaragoza MC, Martinez-Martinez A, Blanco-Lopez MDC, Alegre J. Circulating extracellular vesicles as potential biomarkers in chronic fatigue syndrome/myalgic encephalomyelitis: an exploratory pilot study. J Extracell Vesicles. 2018 Mar 22;7(1):1453730. doi: 10.1080/20013078.2018.1453730. eCollection 2018. PMID 29696075
- [Background] Sotzny F, Blanco J, Capelli E, Castro-Marrero J, Steiner S, Murovska M, Scheibenbogen C; European Network on ME/CFS (EUROMENE). Myalgic Encephalomyelitis/Chronic Fatigue Syndrome - Evidence for an autoimmune disease. Autoimmun Rev. 2018 Jun;17(6):601-609. doi: 10.1016/j.autrev.2018.01.009. Epub 2018 Apr 7. PMID 29635081
- [Background] Scheibenbogen C, Freitag H, Blanco J, Capelli E, Lacerda E, Authier J, Meeus M, Castro Marrero J, Nora-Krukle Z, Oltra E, Strand EB, Shikova E, Sekulic S, Murovska M. The European ME/CFS Biomarker Landscape project: an initiative of the European network EUROMENE. J Transl Med. 2017 Jul 26;15(1):162. doi: 10.1186/s12967-017-1263-z. PMID 28747192
- [Background] Castro-Marrero J, Faro M, Aliste L, Saez-Francas N, Calvo N, Martinez-Martinez A, de Sevilla TF, Alegre J. Comorbidity in Chronic Fatigue Syndrome/Myalgic Encephalomyelitis: A Nationwide Population-Based Cohort Study. Psychosomatics. 2017 Sep-Oct;58(5):533-543. doi: 10.1016/j.psym.2017.04.010. Epub 2017 Apr 21. PMID 28596045
- [Background] Castro-Marrero J, Saez-Francas N, Santillo D, Alegre J. Treatment and management of chronic fatigue syndrome/myalgic encephalomyelitis: all roads lead to Rome. Br J Pharmacol. 2017 Mar;174(5):345-369. doi: 10.1111/bph.13702. Epub 2017 Feb 1. PMID 28052319
- [Background] Castro-Marrero J, Saez-Francas N, Segundo MJ, Calvo N, Faro M, Aliste L, Fernandez de Sevilla T, Alegre J. Effect of coenzyme Q10 plus nicotinamide adenine dinucleotide supplementation on maximum heart rate after exercise testing in chronic fatigue syndrome - A randomized, controlled, double-blind trial. Clin Nutr. 2016 Aug;35(4):826-34. doi: 10.1016/j.clnu.2015.07.010. Epub 2015 Jul 17. PMID 26212172
- [Background] Faro M, Saez-Francas N, Castro-Marrero J, Aliste L, Fernandez de Sevilla T, Alegre J. Gender differences in chronic fatigue syndrome. Reumatol Clin. 2016 Mar-Apr;12(2):72-7. doi: 10.1016/j.reuma.2015.05.007. Epub 2015 Jul 17. English, Spanish. PMID 26190206
- [Background] Castro-Marrero J, Cordero MD, Segundo MJ, Saez-Francas N, Calvo N, Roman-Malo L, Aliste L, Fernandez de Sevilla T, Alegre J. Does oral coenzyme Q10 plus NADH supplementation improve fatigue and biochemical parameters in chronic fatigue syndrome? Antioxid Redox Signal. 2015 Mar 10;22(8):679-85. doi: 10.1089/ars.2014.6181. Epub 2014 Dec 18. PMID 25386668
- [Background] Castro-Marrero J, Cordero MD, Saez-Francas N, Jimenez-Gutierrez C, Aguilar-Montilla FJ, Aliste L, Alegre-Martin J. Could mitochondrial dysfunction be a differentiating marker between chronic fatigue syndrome and fibromyalgia? Antioxid Redox Signal. 2013 Nov 20;19(15):1855-60. doi: 10.1089/ars.2013.5346. Epub 2013 May 29. PMID 23600892
- [Background] Curriu M, Carrillo J, Massanella M, Rigau J, Alegre J, Puig J, Garcia-Quintana AM, Castro-Marrero J, Negredo E, Clotet B, Cabrera C, Blanco J. Screening NK-, B- and T-cell phenotype and function in patients suffering from Chronic Fatigue Syndrome. J Transl Med. 2013 Mar 20;11:68. doi: 10.1186/1479-5876-11-68. PMID 23514202